CLINICAL TRIAL: NCT06259032
Title: Comparative Effect of Mechanical and Functional Alignment in Bilateral Total Knee Arthroplasty on Ankle Alignment : a Randomized Controlled Trial
Brief Title: Comparative Effect of Mechanical and Functional Alignment in Bilateral Total Knee Arthroplasty on Ankle Alignment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 66156
Record Dates: First submitted 2024-01-26; First posted 2024-02-14 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-01

CONDITIONS: Arthropathy of Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mechanical alignment (Experimental)
  Interventions: Other: Mechanical alignment
- Functional alignment (Experimental)
  Interventions: Other: Functional alignment

INTERVENTIONS:
Other: Mechanical alignment — Goal alignment in TKA with mechanical alignment, resection bone in perpendicular to mechanical axis of femur and tibia.
  Arms: Mechanical alignment
Other: Functional alignment — Goal alignment in TKA with functional alignment, resection of bone base on native joint line obliquity.
  Arms: Functional alignment

SUMMARY:
Mechanical alignment (MA) in total knee arthroplasty (TKA) is the most commonly used with well-documented long-term results, however 20% of patients express dissatisfaction following primary TKA. Alternative alignment philosophies have been proposed, aiming to improve patient clinical outcomes and satisfaction. However, evaluation is focused mainly on knee alignment, the pathological findings and other adaptational changes in the ankles and hips are usually neglected.

Thia study aim to comparative effect between mechanical and functional alignment in patient undergone bilateral robotic TKA on ankle alignment and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-80 years
* Symptomatic bilateral knee Osteoarthritis requiring primary TKA
* Willing to undergo bilateral simultaneous TKA
* Able to give informed consent

Exclusion Criteria:

* ligament deficiency requiring constrained prosthesis
* bone loss with augmentation need
* history of fracture around knee or previous osteotomy
* history of ankle fracture
* patient with neuromuscular disorder or movement disorder
* patient is unable to attend the study follow-up program

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Radiographic outcomes : Hip-knee-ankle angle | pre-operative within 2 weeks and post-operative at 2,4,8,12 weeks
  angle in degree between line from center of head of Femur to intercondylar notch and line from tibial interspinous to center of tibial plafond
Radiographic outcomes : Tibial plafond inclination | pre-operative within 2 weeks and post-operative at 2,4,8,12 weeks
  angle in degree between subchondral plate of distal tibial articular surface and vertical axis
Radiographic outcomes :Talar inclination | pre-operative within 2 weeks and post-operative at 2,4,8,12 weeks
  angle in degree between talar dome and vertical axis
Radiographic outcomes : Tibiotalar tilt angle | pre-operative within 2 weeks and post-operative at 2,4,8,12 weeks
  angle in degree between subchondral plate of distal tibial articular surface and talar dome

SECONDARY OUTCOMES:
Clinical outcomes : Knee injury and Osteoarthritis Outcome Score (KOOS) | pre-operative within 2 weeks and post-operative at 2,4,8,12 weeks
  a questionnaire assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.
Clinical outcomes : American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Score | pre-operative within 2 weeks and post-operative at 2,4,8,12 weeks
  evaluation of the clinical status of the ankle-hindfoot, both subjective and objective information. Patients report their pain, and physicians assess alignment. The patient and physician work together to complete the functional portion. Scores range from 0 to 100, with healthy ankles receiving 100 points.
Quality of Life score : EQ-5D-5L | pre-operative within 2 weeks and post-operative at 2,4,8,12 weeks
  assess patient five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels, Index scores range from -0.42 to 1; 1 is the best possible health state. Negative values represent health states perceived as worse than dead, which is equal to 0.
Forgotten Joint Score | pre-operative within 2 weeks and post-operative at 2,4,8,12 weeks
  consists of 12 questions and is transform on a 0-100 scale.The higher the score, the less the patient is aware of their affected joint when performing daily activities

OTHER OUTCOMES:
Other outcomes : soft tissue release | intraoperative
  intra-operative soft tissue release (medial collateral ligament release or others structure around knee) report with Yes (soft tissue release) or No (no soft tissue release)
Other outcomes : operative time | intraoperative
  measured in minutes from skin incision to complete of skin suture
Other outcomes : blood loss | post operative with in 2 days
  record in millilitre measured from Radivac drain
Other outcomes : pain score (Visual analog scale) | post-operative at 2,4,8,12 weeks
  score from 0-10 (0 was no pain, 10 was worst pain )
Other outcomes : Range of knee motion | post-operative at 2,4,8,12 weeks
  record in total degree of knee motion
complications | post-operative at 2,4,8,12 weeks
  Yes (complications) or No ( no complications) if yes, will specified the complications complication such as bone fracture, wound dehiscence, surgical site infection, periprosthetic infection ,pulmonary embolism or other adverse outcomes that may or may not directly associated with the operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No